CLINICAL TRIAL: NCT06455657
Title: Breast Cancer Education for Prisoner Women: Effects on Knowledge and Awareness
Brief Title: Breast Cancer Education to Prisoner Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Principal Investigator, Hitit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Hitit_university_1
Record Dates: First submitted 2024-05-23; First posted 2024-06-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is of a semi-separate type and all women can be trained.
Masking Description: The study is of a semi-separate type and all women can be trained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prisoner women receiving breast cancer training (Experimental): Questionnaires and scales will be administered to the participants as a pre-test. Breast cancer education will be provided in groups and their feedback will be received. Reminder training will be repeated 1 month after the training. The survey and scales will be administered to the participants as a posttest 1 month after the second training.
  Interventions: Other: breast cancer education

INTERVENTIONS:
Other: breast cancer education — Questionnaires and scales will be administered to the participants as a pre-test. Breast cancer education will be provided in groups and their feedback will be received. Reminder training will be repeated 1 month after the training. The survey and scales will be administered to the participants as a posttest 1 month after the second training.

SUMMARY:
this study evaluated the impact of breast cancer education on knowledge and awareness among incarcerated women using a quasi-experimental design.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women in the world, accounting for almost a quarter of cancer cases diagnosed among women, with 1.15 million cases diagnosed each year. Breast cancer is common in both developed and developing countries. However, in developing countries, these rates are three times higher and the mortality rate is quite high. Risk factors include age, low socioeconomic level, early menarche, late menopause, family history of breast disease, long-term use of hormone replacement therapy, breastfeeding status and lifestyle habits.

It is reported that breast cancer screening programs such as mammography, breast self-examination (BSE) and clinical breast examination (CMM) have an important role in early diagnosis, increasing the survival rate, reducing the death rate and preventing relapse in breast cancer patients. It has been reported that women who perform regular BSE are more likely to have early stages of the disease, this is because regular BSE gives the woman information about the feel and appearance of the breast. Thus, the woman will be able to detect any changes as early as possible. It is reported that the practice of breast self-examination depends on different factors, including women's knowledge, attitude, socio-demographic and sociocultural factors. Other reasons for low implementation rates, such as lack of time, forgetfulness, and low education level, have also been reported.

Breast cancer is the second leading cause of death after cervical cancer among incarcerated women under the age of 40. 27% of women over the age of 40 had breast cancer, and 18% of these women died. It is of great importance to raise awareness, which is considered one of the main elements of secondary prevention in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being between the ages of 18-65,
* No history of breast cancer,
* To know Turkish.

Exclusion Criteria:

* Those who do not agree to participate in the study,
* Having a history of breast cancer,
* Those who do not speak Turkish

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Awareness Scale | first-2. months
  The scale is used to measure breast cancer awareness by assessing knowledge of symptoms, appropriate age-related risk, and breast self-examination practices. Higher total scores reflect higher awareness levels.

SECONDARY OUTCOMES:
Comprehensive Breast Cancer Knowledge Test | first- 2. months
  The scale is used to evaluate breast cancer knowledge and perceptions of treatability through true-false statements, with higher scores reflecting greater knowledge levels.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Hitit university, Çorum
  - Fatma Yıldırım, Çorum, Çorum
  - L type prison, Çorum, Çorum

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black E, Richmond R. Improving early detection of breast cancer in sub-Saharan Africa: why mammography may not be the way forward. Global Health. 2019 Jan 8;15(1):3. doi: 10.1186/s12992-018-0446-6. PMID 30621753
- [Background] Choi JS, Park M. Factors predicting young women's willingness to conduct vulvar self-examinations in Korea. Health Care Women Int. 2019 Jun;40(6):653-664. doi: 10.1080/07399332.2018.1531003. Epub 2018 Dec 14. PMID 30550371
- [Background] Jemal A, Bray F, Forman D, O'Brien M, Ferlay J, Center M, Parkin DM. Cancer burden in Africa and opportunities for prevention. Cancer. 2012 Sep 15;118(18):4372-84. doi: 10.1002/cncr.27410. Epub 2012 Jan 17. PMID 22252462
- [Background] Mohamed, A. O. A., Nori, M. M. M., & Altamih, R. A. A. (2021). The Effectiveness of Breast Cancer Health Education Campaign and Breast Self-Examination Training among Female Detainees, Khartoum City-Sudan. Journal of Environmental Science and Public Health, 5(2), 296-310
- [Background] Saadeldin A. Idris, Aamir A. Hamza, Mohamed M. Hafiz, Mohammed Eltayeb A. Ali, Gamal E. H. A., El Shallaly Knowledge, attitude and practice of breast self examination among final years female medical students in Sudan. Int J Public Health Res 2013;1:6-10
- [Result] American Cancer Society. Breast Cancer Information & Overview. 2023. Available from: https://www.cancer.org/cancer/types/breast-cancer.html
- [Result] Baş, S., Ursavaş, F.(2022). Meme Kanseri Farkındalık Ölçeğinin Geçerlilik ve Güvenilirliği, Çankırı Karatekin Üniversitesi Sağlık Bilimleri Enstitüsü Hemşirelik Anabilim Dalı, Yüksek Lisans Tezi